CLINICAL TRIAL: NCT01472939
Title: A Phase 2b, Double-blind, Randomized, Placebo-controlled, Dose-finding Study to Evaluate Efficacy of a Selective 5-HT4 Receptor Agonist and Proton Pump Inhibitor (PPI) in Subjects With Gastroesophageal Reflux Disease (GERD) With Persistent Regurgitation With or Without Heartburn
Brief Title: Selective 5-HT4 Receptor Agonist and Proton Pump Inhibitor (PPI) in Subjects With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD557-206; 2011-004388-62 (EudraCT Number)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — revexepride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SSP-002358 (0.1 mg) + Proton Pump Inhibitor (PPI) (Active Comparator)
  Interventions: Drug: SSP-002358 (0.1 mg) + PPI
- SSP-002358 (0.5 mg) + PPI (Active Comparator)
  Interventions: Drug: SSP-002358 (0.5 mg) + PPI
- SSP-002358 (2.0 mg) + PPI (Active Comparator)
  Interventions: Drug: SSP-002358 (2.0 mg) + PPI
- Placebo + PPI (Placebo Comparator)
  Interventions: Drug: Placebo + PPI

INTERVENTIONS:
Drug: SSP-002358 (0.1 mg) + PPI — 0.1 mg tablet three times daily (t.i.d.) taken in addition to a PPI
  Other Names: SPD557
  Arms: SSP-002358 (0.1 mg) + Proton Pump Inhibitor (PPI)
Drug: SSP-002358 (0.5 mg) + PPI — 0.5 mg tablet t.i.d. taken in addition to a PPI
  Arms: SSP-002358 (0.5 mg) + PPI
Drug: SSP-002358 (2.0 mg) + PPI — 2.0 mg tablet t.i.d. taken in addition to a PPI
  Arms: SSP-002358 (2.0 mg) + PPI
Drug: Placebo + PPI — Placebo t.i.d. taken in addition to a PPI
  Arms: Placebo + PPI

SUMMARY:
The aim of this study is to establish a dose-related effect of a selective 5-HT4 receptor agonist compared to placebo on residual symptoms (regurgitation with or without heartburn) in subjects with GERD who have persistent symptoms while on PPI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent Form signed voluntarily before the first study-related activity.
2. Aged between 18 and 70 years, inclusive.
3. Subjects with a history of the cardinal symptoms of GERD (both heartburn and regurgitation) prior to PPI therapy.
4. Subjects with symptoms of GERD for at least 6 months prior to the Screening Visit.
5. Subjects who have persistent symptoms of regurgitation for 3 or more days over the past week with or without heartburn while on PPI.
6. Subjects have at least some improvement to the symptom of heartburn while on PPI therapy.
7. Subjects on PPI therapy for at least 8 weeks prior to the Screening Visit of which the last 4 weeks are on a stable labeled dose for any GERD indication according to the country label, where a change of PPI therapy would not impact the symptoms (twice-daily dosing of PPI is not allowed in the last 4 weeks)

Exclusion Criteria:

1. Subjects who show no response to heartburn while on PPI therapy.
2. Subjects with dyspepsia symptoms that are more predominant than their GERD symptoms (heartburn and/or regurgitation).
3. Subjects with prior endoscopic anti-reflux procedure or major GI surgery or subjects with major GI disorders.
4. Presence of severe and clinically uncontrolled cardiovascular, liver, lung or neurologic disease, cancer or AIDS.
5. Alarm symptoms suggestive of malignancies or organic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2013-05-14 (Actual); Study Completion 2013-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (88):
- United States (62):
  - HOPE Research Institute, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Southern California Research Institute Medical Group Inc, Los Angeles, California
  - Medical Center for Clinical Research, San Diego, California
  - Clinicos, Colorado Springs, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Medical Research Unlimited, LLC, Aventura, Florida
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - PAB Clinical Research, Brandon, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Medical Research Unlimited, LLC, Hialeah, Florida
  - Jupiter Research, Jupiter, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Radiant Research, Pinellas Park, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Gastrointestinal Specialists of GA, PC, Marietta, Georgia
  - Digestive Research Associates, Newnan, Georgia
  - Rockford Gastroenterology Associates, Ltd, Rockford, Illinois
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Research Integrity, Owensboro, Kentucky
  - Clinical Trials Management, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Meritus Medical Center, Hagerstown, Maryland
  - Beacon Clinical Research, Brockton, Massachusetts
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - New Jersey Physicians, LLC, Clifton, New Jersey
  - UNC Hospitals, Chapel Hill, North Carolina
  - Carolinas Research Associates, Davidson, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Vital Research, Inc., Greensboro, North Carolina
  - Carolinas Research Associates, Harrisburg, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - Oklahoma Foundation for Digestive Research Sciences Center, Oklahoma City, Oklahoma
  - Family Medical Associates, Levittown, Pennsylvania
  - Guthrie Clinic, Ltd., Sayre, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Clinsearch, LLC, Chattanooga, Tennessee
  - Radiant Research Dallas-North, Dallas, Texas
  - GI Consultants, P.A., Houston, Texas
  - Pasadena Gastroenterology Assoc, dba Digestive Health Center, Pasadena, Texas
  - Office Based Practitioner, San Antonio, Texas
  - Advanced Research Institute, Clinton, Utah
  - Advanced Research Institute, Logan, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute, Sandy City, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Blue Ridge Medical Center, Lynchburg, Virginia
  - Ramstad Medical Associates, Suffolk, Virginia
  - Aurora Wilkinson Medical Clinic, Summit, Wisconsin
- Czechia (2):
  - Hepato-Gastroenterology HK s.r.o., Hradec Králové
  - Nemocnice Valasske Mezirici a.s., Valašské Meziříčí
- Germany (7):
  - Praxis Dr. Andreas Schwittay-Facharzt fuer Innere Medizin, Böhlen
  - Zentrum fur Innere Medizin, Klinikum Garmisch Partenkirchen, Garmisch-Partenkirchen
  - Haus der Gesundheit, Ludwigshafen
  - Praxis für Gastroenterologie und fachärztliche Innere Medizin, Ludwigshafen
  - Medizinische Fakultät der Otto-von-Guericke Universität, Magdeburg
  - Gemeinschaftspraxis Dres. Brandt, Potsdam
  - Gemeinschaftspraxis Dres Josef und Wilma Großkopf, Wallerfing
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Pauls Stradins Clinical University Hospital, Riga
  - Digestive Disease Centre "Gastro", Riga
  - Vidzemes Hospital, Valmiera
- Poland (9):
  - NZOZ Specjalistyczne Centrum Gastrologii Gastromed, Bialystok
  - Centrum Medyczne im Swietego Lukasza Sp. z o.o., Częstochowa
  - NZOZ ''Salvia'', Katowice
  - Centrum Medyczne Szpital sw. Rodziny Sp. z o.o., Lodz
  - Gastromed Sp. K. NZOZ, Lublin
  - Endoskopia Sp. z o.o., Sopot
  - NZOZ Vivamed, Warsaw
  - Lexmedica, Wroclaw
  - Aktywne Centrum Zdrowia NZOZ ZAWIDAWIE Sp. z o.o., Wroclaw
- Romania (4):
  - Brasov County Hospital, Brasov
  - Centrul Medical Galenus, Târgu Mureş
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
  - Policlinica "Dr. Citu" SRL, Timișoara

REFERENCES:
- [Derived] Shaheen NJ, Adler J, Dedrie S, Johnson D, Malfertheiner P, Miner P, Meulemans A, Poole L, Tack J, Thielemans L, Troy S, Vakil N, Zerbib F, Ruth M. Randomised clinical trial: the 5-HT4 agonist revexepride in patients with gastro-oesophageal reflux disease who have persistent symptoms despite PPI therapy. Aliment Pharmacol Ther. 2015 Apr;41(7):649-61. doi: 10.1111/apt.13115. Epub 2015 Feb 19. PMID 25693609

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + PPI: Placebo taken three times daily (TID) in addition to a PPI
- SSP-002358 0.1mg + PPI: 0.1 mg tablet taken TID in addition to a PPI
- SSP-002358 0.5mg + PPI: 0.5 mg tablet taken TID in addition to a PPI
- SSP-002358 2.0mg + PPI: 2.0 mg tablet taken TID in addition to a PPI
Period: Overall Study
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Started | 123 | 119 | 119 | 119
Completed | 103 | 105 | 108 | 99
Not Completed | 20 | 14 | 11 | 20
Not completed — Adverse Event | 3 | 7 | 7 | 14
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 0 | 2 | 0
Not completed — Clinically Significant Pre-Dose ECG | 0 | 0 | 1 | 0
Not completed — Prohibited Medication | 0 | 1 | 0 | 0
Not completed — Withdrawal By PI | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set was used which consisted of all randomized subjects who took at least 1 dose of investigational product. Three subjects did not receive investigational product, therefore n=477.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI | Total
Number analyzed (Participants) | 122 | 119 | 118 | 118 | 477
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (12.1) | 48.8 (12.59) | 49.2 (12.31) | 47.6 (11.3) | 47.9 (12.11)
Age, Customized [Count of Participants; unit: Participants]
  18 - 40 | 40 | 35 | 29 | 32 | 136
  41 - 50 | 35 | 23 | 32 | 32 | 122
  51 - 65 | 41 | 52 | 49 | 51 | 193
  >65 | 6 | 9 | 8 | 3 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 72 | 65 | 289
  Male | 48 | 41 | 46 | 53 | 188
Region of Enrollment [Count of Participants; unit: Participants] — All randomized subjects (n = 480)
  Participants
    CZECH REPUBLIC | 1 | 1 | 1 | 1 | 4
    FRANCE | 2 | 2 | 1 | 2 | 7
    GERMANY | 5 | 4 | 4 | 4 | 17
    HUNGARY | 3 | 1 | 2 | 1 | 7
    LATVIA | 5 | 4 | 4 | 4 | 17
    POLAND | 6 | 7 | 7 | 8 | 28
    ROMANIA | 9 | 8 | 8 | 8 | 33
    UNITED STATES | 92 | 92 | 92 | 91 | 367

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Regurgitation-Free Days Over Weeks 5-8
Time Frame: Baseline and over weeks 5-8
Population: Full Analysis Set consisted of all subjects in the Safety Analysis Set who had at least 1 post-baseline value for the primary efficacy assessment. Safety Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 120 | 119 | 114 | 113
percentage of days | 36.96 (3.598) | 43.01 (3.678) | 44.37 (3.667) | 38.79 (3.728)
Statistical Analysis 1: Comparison: Placebo + PPI vs SSP-002358 0.1mg + PPI; Test type: Superiority or Other; p = 0.128, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 6.06, 95% CI 2-sided [-1.743 to 13.862]
Statistical Analysis 2: Comparison: Placebo + PPI vs SSP-002358 0.5mg + PPI; Test type: Superiority or Other; p = 0.062, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 7.42, 95% CI 2-sided [-0.378 to 15.212]
Statistical Analysis 3: Comparison: Placebo + PPI vs SSP-002358 2.0mg + PPI; Test type: Superiority or Other; p = 0.650, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 1.83, 95% CI 2-sided [-6.100 to 9.765]

2. Secondary Outcome: Change From Baseline in Heartburn-Free Days Over Weeks 5-8
Time Frame: Baseline and over weeks 5-8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 120 | 119 | 114 | 113
percentage of days | 21.76 (3.623) | 28.52 (3.686) | 30.68 (3.688) | 27.47 (3.756)
Statistical Analysis 1: Comparison: Placebo + PPI vs SSP-002358 0.1mg + PPI; Test type: Superiority or Other; p = 0.102, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 6.75, 95% CI 2-sided [-1.344 to 14.850]
Statistical Analysis 2: Comparison: Placebo + PPI vs SSP-002358 0.5mg + PPI; Test type: Superiority or Other; p = 0.031, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 8.92, 95% CI 2-sided [0.814 to 17.021]
Statistical Analysis 3: Comparison: Placebo + PPI vs SSP-002358 2.0mg + PPI; Test type: Superiority or Other; p = 0.175, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = 5.71, 95% CI 2-sided [-2.540 to 13.957]

3. Secondary Outcome: Change From Baseline in the Persistent Reflux Integrated Symptom Measurement (PRISM) Liquid and Food Domain Scores Over Weeks 5-8
Description: PRISM is a 21 item patient-reported outcome instrument with 4 domains. Items are scored using various scales. Total score ranges from 0-100. Higher scores indicate more severe or frequent symptoms.
Time Frame: Baseline and over weeks 5-8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 120 | 119 | 114 | 113
units on a scale | -13.29 (1.206) | -15.77 (1.228) | -16.49 (1.235) | -15.44 (1.250)
Statistical Analysis 1: Comparison: Placebo + PPI vs SSP-002358 0.1mg + PPI; Test type: Superiority or Other; p = 0.064, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-5.087 to 0.141]
Statistical Analysis 2: Comparison: Placebo + PPI vs SSP-002358 0.5mg + PPI; Test type: Superiority or Other; p = 0.017, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-5.818 to -0.573]
Statistical Analysis 3: Comparison: Placebo + PPI vs SSP-002358 2.0mg + PPI; Test type: Superiority or Other; p = 0.114, Mixed Models Repeated Measures Analysis; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-4.813 to 0.519]

4. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUC) of SSP-002358
Description: Area under the plasma concentration versus time curve can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 8 hours post-dose (week 2 or later)
Population: Full Pharmacokinetic Subset consisted of a subset of subjects who underwent the detailed pharmacokinetic assessments. Subjects who vomited within the blood sampling period may have been excluded.
Measure: Mean (Standard Deviation); unit: pg*h/ml
Arm/Group | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 12 | 9 | 8
pg*h/ml | 1650 (729) | 8352 (2564) | 42613 (4971)

5. Secondary Outcome: Steady State Maximum Plasma Concentration (Cmax) of SSP-002358
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administered.
Time Frame: Over 8 hours post-dose (week 2 or later)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 12 | 9 | 8
pg/ml | 648 (302) | 3374 (1175) | 17900 (3573)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of SSP-002358
Time Frame: Over 8 hours post-dose (week 2 or later)
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Number analyzed (Participants) | 12 | 9 | 8
hours | 5.00 [0.483 to 5.58] | 5.07 [5.00 to 5.55] | 4.51 [1.00 to 5.48]

ADVERSE EVENTS:
Description: Safety Analysis Set consisted of all randomized subjects who took at least 1 dose of investigational product (n = 477).
Arm/Group | Placebo + PPI | SSP-002358 0.1mg + PPI | SSP-002358 0.5mg + PPI | SSP-002358 2.0mg + PPI
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/119 | 0/118 | 1/118
Other Adverse Events (participants affected / at risk) | 25/122 | 22/119 | 35/118 | 45/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + PPI (N=122) | SSP-002358 0.1mg + PPI (N=119) | SSP-002358 0.5mg + PPI (N=118) | SSP-002358 2.0mg + PPI (N=118)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + PPI (N=122) | SSP-002358 0.1mg + PPI (N=119) | SSP-002358 0.5mg + PPI (N=118) | SSP-002358 2.0mg + PPI (N=118)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 12 (12) | 19 (20) | 32 (33)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (7) | 5 (5) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4) | 7 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 7 (7) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.